CLINICAL TRIAL: NCT05117151
Title: Ability of Hypotension Prediction Index to Predict Future Hypotension Events in Each Phase of Thoracic Surgery: an Observational Pilot Study
Brief Title: Ability of Hypotension Prediction Index to Predict Hypotension Events in Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202109061RIND
Record Dates: First submitted 2021-10-31; First posted 2021-11-11 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Perioperative/Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observation: monitor intraoperative hypotension prediction index as well as hemodynamic variables to exam the ability in predicting hypotension events of each variable
  Interventions: Diagnostic Test: hypotension prediction index

INTERVENTIONS:
Diagnostic Test: hypotension prediction index — monitor intraoperative hypotension prediction index as well as hemodynamic variables to exam the ability in predicting hypotension events of each variable

SUMMARY:
Investigators design this prospective observational study to exam the ability of hypotension prediction index in predicting intraoperative hypotension events in each phase of thoracic surgery

DETAILED DESCRIPTION:
Hypotension prediction index is a novel introduced monitoring-tool that aims to predict hypotension events before their occurence, and has been reported to have superior predictive ability than the commonly measured perioperative hemodynamic variables. To date, there is no information regarding its ability to predict hypotension events in each phase of thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* adults undergoing scheduled VATS surgery

Exclusion Criteria:

* pregnant women
* patients in intensive care units
* patients with the underlying disease including respiratory failure(FEV1/FVC < 70 % and FEV1 < 50%), heart failure(NYHA score =III、IV), kidney failure(eGFR< 60 ml.min-1.1.73m-2), liver failure
* patients with ongoing infection

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults undergoing scheduled VATS surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
ability of hypotension prediction index in predicting hypotension events | 3 hours
  to calculate the sensitivity/specificity and AUROC of hypotension prediction index in predicting hypotension events

SECONDARY OUTCOMES:
ability of dynamic parameters in predicting hypotension events | 3 hours
  to calculate the sensitivity/specificity and AUROC of dynamic parameters in predicting hypotension events

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Yu Wu, Ph.D., Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Monk TG, Bronsert MR, Henderson WG, Mangione MP, Sum-Ping ST, Bentt DR, Nguyen JD, Richman JS, Meguid RA, Hammermeister KE. Association between Intraoperative Hypotension and Hypertension and 30-day Postoperative Mortality in Noncardiac Surgery. Anesthesiology. 2015 Aug;123(2):307-19. doi: 10.1097/ALN.0000000000000756. PMID 26083768
- [Background] Hatib F, Jian Z, Buddi S, Lee C, Settels J, Sibert K, Rinehart J, Cannesson M. Machine-learning Algorithm to Predict Hypotension Based on High-fidelity Arterial Pressure Waveform Analysis. Anesthesiology. 2018 Oct;129(4):663-674. doi: 10.1097/ALN.0000000000002300. PMID 29894315
- [Background] Wijnberge M, Geerts BF, Hol L, Lemmers N, Mulder MP, Berge P, Schenk J, Terwindt LE, Hollmann MW, Vlaar AP, Veelo DP. Effect of a Machine Learning-Derived Early Warning System for Intraoperative Hypotension vs Standard Care on Depth and Duration of Intraoperative Hypotension During Elective Noncardiac Surgery: The HYPE Randomized Clinical Trial. JAMA. 2020 Mar 17;323(11):1052-1060. doi: 10.1001/jama.2020.0592. PMID 32065827